CLINICAL TRIAL: NCT05459597
Title: Population Pharmacokinetics, Effectiveness and Safety of Antiepileptic Drugs in Elderly Patients
Brief Title: Antiepileptic Drugs in Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Wei Zhao (Other)
Collaborators: Qianfoshan Hospital (Other); The Second Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor-Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Organization: Shandong University (Other)
Other Study IDs: Elderly-Antiepileptic Drugs
Record Dates: First submitted 2022-07-04; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Seizure, Epileptic
MeSH Terms: conditions — Seizures | interventions — Anticonvulsants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: The use of antiepileptic drugs depends on the clinical practice.
  Interventions: Drug: antiepileptic drugs

INTERVENTIONS:
Drug: antiepileptic drugs — phenytoin, carbamazepine, lamotrigine, levetiracetam, perampanel, etc. as part of routine treatment.

SUMMARY:
The purpose is to study the population pharmacokinetics, effectiveness and safety of antiepileptic drug (phenytoin, carbamazepine, lamotrigine, levetiracetam, parempanel, etc) in elderly patients and recommend optimized dosage regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years old;
2. Diagnosed with epilepsy;
3. Using antiepileptic drugs for treatment;

Exclusion Criteria:

1. Patients who are expected to die within 48 hours;
2. Patients with allergy to antiepileptic drugs;
3. Patients receiving other investigational drugs;
4. Other factors that the researcher considers unsuitable for inclusion.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with epilepsy (≥65years).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The peak plasma drug concentration of antiepileptic drugs. | at (0-4) h after oral administration
  To detect the peak plasma drug concentration of antiepileptic drugs.
The random plasma drug concentration of antiepileptic drugs. | at (4-10) h after oral administration
  To detect the random plasma drug concentration of antiepileptic drugs.
The trough plasma drug concentration of antiepileptic drugs. | at (1-2) h before the next administration
  To detect the trough plasma drug concentration of antiepileptic drugs.

SECONDARY OUTCOMES:
The incidence of adverse drug reaction | Through study completion, an average of 14 days
The frequency of seizures | Through study completion, an average of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Study Chair — Qianfoshan Hospital
Locations (1):
- Wei Zhao, Jinan, Shandong, China